CLINICAL TRIAL: NCT03590717
Title: Impact Evaluation of WFP's Fresh Food Voucher Pilot Programme in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: Addis Ababa University (Other); United Nations World Food Programme (WFP) (Other)
Responsible Party: Principal Investigator, Kalle Hirvonen, Research Fellow, International Food Policy Research Institute
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 699013
Record Dates: First submitted 2018-07-06; First posted 2018-07-18 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Diet; Deficiency; Malnutrition
Keywords: dietary diversity; minimum acceptable diet; fruits; vegetables; animal sourced foods
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial clustered at the village level, 2 treatment arms and one control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BCC-Only (Other): Intervention: Households in the 'BCC-only' arm receive SBCC but do not receive vouchers.
  Interventions: Behavioral: BCC-Only
- Small-voucher (Experimental): Intervention: Households in the 'Small-voucher' arm receive a voucher (~$12-17) every month that entitles them to purchase fresh foods (fruits, vegetables and animal sourced foods). The households in this arm also receive the same social behavioural change communication (SBCC) messages as the 'BCC-only' arm.
  Interventions: Other: Small-voucher
- Large-voucher (Experimental): Intervention: Households in the 'Large-voucher' arm receive a larger voucher (~$21-23) every month that entitles them to purchase fresh foods (fruits, vegetables and animal sourced foods). The households in this arm also receive the same social behavioural change communication (SBCC) messages as the 'BCC-only' arm.
  Interventions: Other: Large-voucher

INTERVENTIONS:
Behavioral: BCC-Only — Households in the 'BCC-only' arm receive SBCC but do not receive vouchers.
  Arms: BCC-Only
Other: Small-voucher — Households in the 'Small-voucher' arm receive a voucher (~$12-17) every month that entitles them to purchase fresh foods (fruits, vegetables and animal sourced foods). The households in this arm also receive the same social behavioural change communication (SBCC) messages as the 'BCC-only' arm.
  Arms: Small-voucher
Other: Large-voucher — Households in the 'Large-voucher' arm receive a larger voucher (~$21-23) every month that entitles them to purchase fresh foods (fruits, vegetables and animal sourced foods). The households in this arm also receive the same social behavioural change communication (SBCC) messages as the 'BCC-only' arm.
  Arms: Large-voucher

SUMMARY:
To assess the impact of WFP's Fresh Food Voucher Pilot Programme in Ethiopia on children's and mother's diets

DETAILED DESCRIPTION:
Rationale: Infants, young children and adult women in rural Ethiopia consume one of the least diversified diets in the world. The World Food Programme's Fresh Food Voucher (FFV) Pilot Programme aims to improve dietary diversity among infants and young children and their mothers. The focus on these demographic groups is based on the now well-established theory on the importance of the 'first 1,000 days'. This period, spanning the pregnancy and the first 2 years of child's life, is considered critical for child's physical growth and cognitive development. The beneficiary households receive a voucher that can be used to purchase fresh foods (fruits, vegetables and certain animal source foods).

Objective: The main objectives of the evaluation are to assess and report on the performance and results of the FFV programme to help WFP present high-quality and credible evidence of actual impact to its donors. In addition, the evaluation will determine the reasons why certain results occurred (or not) to draw lessons, derive good practices and pointers for learning.

Study design: This is a mixed methods evaluation that combines a Randomized Controlled Trial (RCT) with Focus Group Discussions (FGDs) with caregivers and food traders. The RCT contains three arms. The first treatment arm receives a smaller voucher (roughly $12-17) and social behavioural change communication (SBCC). The second treatment arm receives a larger voucher (roughly $21-23) and SBCC. Households in the third study arm (control) receive SBCC but do not receive vouchers. A cluster in this impact evaluation is defined as a village (got in Amharic) and these clusters of are randomly allocated to the different arms of the trial. Within a cluster, all eligible households will receive the same treatment.

Study population: All households with a child between 6-17 months at the baseline in December 2017 were eligible to be included in the quantitative sample.

Main study parameters/endpoints: The main outcomes of interest are minimum acceptable diet score for children 6- 23 months (World Health Organization, 2008) and minimum diet diversity for women of reproductive age (FAO & FHI-360, 2016).

ELIGIBILITY:
Inclusion Criteria:

Households with young children aged 6-17 months age at the baseline in December 2017.

Ages: 6 Months to 17 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 574 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Minimum Acceptable Diet Scores (MAD) of children 6-23 months of age | 12 months
  Change in the proportion of children achieving MAD
Minimum diet diversity (MDD-W) for women of reproductive age | 12 months
  Change in the proportion of women achieving MDD-W

SECONDARY OUTCOMES:
Minimum Diet Diversity (MDD) of children 6-23 months of age | 12 months
  Change in the proportion of children achieving MDD
Minimum Meal Frequency (MFF) of children 6-23 months of age | 12 months
  Change in the proportion of children achieving MFF
Household Diet Diversity Score (HDDS) | 12 months
  Mean difference in HDDS
WFP Food Consumption Score- Nutrition | 12 months
  Mean difference in WFP Food Consumption Score- Nutrition

CONTACTS AND LOCATIONS:
Overall Officials: Kalle Hirvonen, PhD, Principal Investigator — International Food Policy Research Institute, Ethiopia; Kaleab Baye, PhD, Principal Investigator — Center for Food Science and Nutrition, Addis Ababa University, Ethiopia
Locations (1):
- Kalle Hirvonen, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided